CLINICAL TRIAL: NCT06725836
Title: Clinical Testing and Assessment of the Physiological Effects of Invasive Spinal Cord Stimulation Using Electroencephalography to Optimize Rehabilitation Programs and Develop Personalized Approaches for Recovery After Spinal Injury
Brief Title: Clinical Testing of Invasive Spinal Cord Stimulation and Evaluation of Its Physiological Effects Using the Electroencephalography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artur Biktimirov (Other)
Collaborators: Skolkovo Institute of Science and Technology (Other); The Federal Center of Brain Research and Neurotechnologies (Unknown)
Responsible Party: Sponsor-Investigator, Artur Biktimirov, Head of the Laboratory of Experimental and Translational Medicine of Far Eastern Federal University (FEFU), Far Eastern Federal University
Organization: Far Eastern Federal University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DVFU-04
Record Dates: First submitted 2024-12-04; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries (SCI); Spinal Cord Injury
Keywords: Spinal Cord Stimulation; Electric Stimulation Therapy; Spinal Cord Injuries; Rehabilitation; Brain Waves; Central Nervous System; EEG
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spinal Cord Stimulation (Experimental): Patients with clinical presentations of complete and incomplete spinal cord injury.
  Interventions: Procedure: Implantation of electrodes into the epidural space for spinal cord stimulation; Procedure: Selection of the optimal spinal cord stimulation program for spastic syndrome suppression; Procedure: Selection of the optimal spinal cord stimulation program for volitional motor control; Diagnostic Test: Resting electroencephalography for identifying neurocorrelates of spinal cord stimulation.; Diagnostic Test: Electroencephalography within the motor imagery paradigm

INTERVENTIONS:
Procedure: Implantation of electrodes into the epidural space for spinal cord stimulation — Under X-ray guidance and with neurophysiological supervision, the electrode is implanted. The stimulator is surgically placed in a pocket formed in the iliac crest area on the left side, where it is secured. The generator is connected to an electrode array positioned on the dorsal epidural surface of the spinal cord at the appropriate level (sacral-lumbar/cervical region), as confirmed by intraoperative fluoroscopy.
Procedure: Selection of the optimal spinal cord stimulation program for spastic syndrome suppression — During the selection of the optimal stimulation program for spasticity suppression, spinal cord stimulation (SCS) is performed at various sites on the electrode array. Stimulation is initiated at a specific site with a frequency of 60 Hz, and the intensity is gradually increased until the spasticity is alleviated (i.e., the limb can flex and extend without restriction). If there is no effect, the stimulation frequency is increased by 5 Hz, and the intensity is again adjusted from 0 to comfortable values. Stimulation is sequentially applied at different sites, and those sites where muscle spasticity is most effectively suppressed are selected.
Procedure: Selection of the optimal spinal cord stimulation program for volitional motor control — Over the course of two weeks, the configuration of the electrodes and the intensity of the stimulation are adjusted to ensure optimal voluntary muscle control. A systematic approach is used to determine the most suitable settings. First, the anodes and cathodes on the electrode array are identified. The desired frequency range is 20-40 Hz. The pulse width is determined empirically. The adjustment begins at 20 Hz, with the stimulation intensity gradually increased. If unpleasant sensations (such as muscle spasms or pain) occur, the intensity is reduced to comfortable values. If there is no effect, the stimulation frequency is increased by 5 Hz, and the intensity is adjusted again from 0 to comfortable levels. Stimulation is sequentially applied at different sites, with the sites that provide the most effective voluntary muscle control being selected.
Diagnostic Test: Resting electroencephalography for identifying neurocorrelates of spinal cord stimulation. — The procedure utilizes the method of electroencephalography (EEG). Throughout the procedure, EEG signals are recorded. Initially, the participant is recorded in a resting state before the implantation of the stimulator for 20 minutes (5 minutes with eyes open, followed by 5 minutes with eyes closed). After the surgery, the participant is recorded in the same manner before the first activation of the stimulator. After selecting the programs, the participant is recorded without stimulation (eyes open, then closed), followed by recordings with the spinal cord stimulator (SCS) activated (eyes open, then closed). The stimulation is then turned off again, and recording is conducted with eyes open and closed. Before discharge, the participant is recorded in a resting state for 20 minutes with the stimulation program active.
Diagnostic Test: Electroencephalography within the motor imagery paradigm — The procedure utilizes the method of electroencephalography (EEG). Throughout the procedure, EEG signals are recorded. During the experiment, with the stimulator turned off, the participant views a fixation cross on a computer screen. Then, they hear an auditory signal and see a sign indicating a specific movement (complete flexion and extension of the left arm, complete flexion and extension of the right arm, complete flexion and extension of the left leg, complete flexion and extension of the right leg). The participant imagines the movements according to the auditory and visual signals on the screen. Subsequently, the participant performs the same movements in the same order. The motor control stimulation program is then activated, and the entire sequence is repeated (first imagining the movement, then performing the imagined movements). The timing of the command presentations is recorded with marker placements.

SUMMARY:
The aim of the study is to identify the specific characteristics of brain network dysfunctions and assess the recovery of their functionality through the recording of resting-state electroencephalography (EEG) during rehabilitation using spinal cord stimulation (SCS). Researchers expect that effective SCS scenarios will result in progressive alterations in the quantitative metrics of resting-state EEG throughout the rehabilitation period. The data obtained may be used to optimize rehabilitation protocols and develop personalized approaches for recovery after spinal cord injury.

DETAILED DESCRIPTION:
The aim of the study is to identify the nature of brain network dysfunctions and assess the recovery of their function based on resting-state electroencephalography (EEG) recordings during rehabilitation using spinal cord stimulation (SCS).

The study aims to gather information on the role of brain neuroplasticity during the use of effective SCS programs with implanted electrodes in participants with partial or complete spinal cord injury at various levels.

Participants are enrolled according to inclusion criteria. Before the procedure for implanting multichannel electrodes, resting-state EEG recordings are performed. Then, multichannel electrodes are implanted into the epidural space of the spinal cord below the level of injury. After the implantation, another resting-state EEG recording is conducted before the stimulator is turned on for the first time. Once the optimal SCS program is selected (for the suppression of spastic syndrome or volitional motor control), periodic resting-state EEG recordings are made: before stimulation, during stimulation, and after stimulation. Before the participant is discharged, a final resting-state EEG recording is performed with the stimulator turned on. Scheduled postoperative monitoring will be conducted for up to 2 weeks.

SCS is initiated on the second day after the surgical procedure. The participant is instructed on the use of the stimulator. The optimal program is selected within commonly accepted ranges of stimulation parameters (frequency, amplitude, pulse width) based on maximum efficacy.

Researchers expect that effective SCS scenarios will result in progressive alterations in the quantitative metrics of resting-state EEG throughout the rehabilitation period. The data obtained may be used to optimize rehabilitation protocols and develop personalized approaches for recovery after spinal cord injury.

Within the motor imagery paradigm, following the selection of the program for volitional motor control, participants are instructed to sequentially imagine movements of the limbs (general flexion and extension of the left arm, general flexion and extension of the right arm, general flexion and extension of the left leg, and general flexion and extension of the right leg) in response to auditory and visual cues displayed on a computer screen. After imagining these movements, participants are required to physically perform the same movements. Recordings are made with the stimulator both turned off and on. Throughout the entire recording period, EEG is continuously recorded from the participant. The primary aim of this recording is to investigate the desynchronization of the mu rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with implanted spinal cord stimulation device
* Patients undergoing a scheduled implantation of a spinal cord stimulation device
* Complete spinal cord injury
* Incomplete spinal cord injury

Exclusion Criteria:

* Presence of severe somatic pathology that prevents surgical treatment and participation in the study
* Presence of mental disorders, severe depression, or a history of suicidal tendencies
* History of oncology
* History of epilepsy
* History of stroke
* Inability to perform electrical stimulation due to other somatic pathology
* Purulent-septic pathology
* Drug addiction (including in the medical history)
* Central nervous system developmental anomalies
* Any conditions that, in the investigator's opinion, meet the exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-04-22 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Spectral characteristics of resting electroencephalography in standard frequency bands during neurostimulator turned on/off and with eyes open/closed | Up to 2 weeks
  Electroencephalography (EEG) spectral power in standard frequency bands (1-40 Hz) will be analyzed across different conditions: stimulator on vs. off, and eyes open vs. closed. Independent component analysis (ICA) will be used for artifact removal, followed by spectral power computation and normalization.
Spatial distribution of electroencephalography rhythms in standard frequency bands during neurostimulator turned on/off and with eyes open/closed | Up to 2 weeks
  This outcome evaluates the spatial patterns of electroencephalography (EEG) rhythms across the scalp in standard frequency bands. Independent component analysis (ICA) will correct artifacts, and spatial maps of EEG power will be compared between the neurostimulation conditions (on/off) and different visual states (eyes open/closed). This analysis will help identify brain regions influenced by SCS.
Functional connectivity measures in standard frequency bands (imaginary part of coherence, PLV, etc.) during neurostimulation on/off and with eyes open/closed | Up to 2 weeks
  Functional connectivity between brain regions will be measured using metrics such as coherence and phase-locking value (PLV) in standard frequency bands. The analysis will focus on how connectivity patterns change with the stimulator on vs. off and eyes open vs. closed, providing insights into network-level effects of spinal cord stimulation.
Mu rhythm desynchronization within the motor imagery paradigm during neurostimulation on/off and with eyes open/closed | Up to 2 weeks
  Changes in mu rhythm desynchronization during motor imagery will be evaluated as a marker of motor cortex engagement. Electroencephalography (EEG) will be recorded during imagined limb movements, with and without neurostimulation. The comparison will determine the effect of spinal cord stimulation (SCS) on motor-related brain activity.

SECONDARY OUTCOMES:
American Spine Injury Association / International Standards for Neurological and Functional Classification of Spinal Cord Injury (ASIA/ISCSCI) | Baseline
  The ASIA/ISNCSCI is a standardized quantitative system for assessing the neurological status of patients with spinal cord injuries. The assessment algorithm involves sequential determination of the following: sensory levels of injury on the right and left sides by dermatome (where 0 - absent, 1 - impaired/altered sensation (reduced or hypersensitivity), and 2 - normal sensation); motor levels of injury on the right and left sides (ranging from 0, which represents complete paralysis, to 5, which represents normal active movement); the neurological level of injury; completeness of injury (complete or incomplete); and the degree of spinal cord injury (A - complete injury; B - complete absence of motor function but with preserved sensation; C - significant motor function impairment with preserved sensation; D - mild motor impairments with normal sensation and functionally significant movements; E - sensation and motor function are graded as normal).
The Short Form-36 (SF-36) | Baseline
  The Short Form-36 consists of eight scales: physical functioning, physical role functioning, bodily pain, general health perceptions, vitality, social role functioning, emotional role function, and mental health. Each scale ranges from 0 (worst possible score) to 100 (best possible score).
Spinal Cord Independence Measure III (SCIM-III) | Baseline
  The SCIM-III scale consists of three subscales: self-care (eating, bathing, dressing), respiration and sphincter management, and mobility (in bed and transfers in/out of the room). The results are determined by summing the points of all items, yielding a total score (ranging from 0 to 100) and/or by summing the subscale scores (self-care: 0-20; respiration and sphincter management: 0-40; mobility: 0-40).
The Neurogenic Bladder Symptom Score (NBSS) | Baseline
  The NBSS scale allows for the assessment of symptom severity regardless of the type of neurogenic dysfunction and whether or not the patient has voluntary urination. The scale consists of 24 items that measure bladder symptoms across 3 different domains: incontinence (ranging from 0 to 29), storage and voiding (from 0 to 22), and consequences (from 0 to 23). There is also a single general question about quality of life related to urination, rated on a scale from 0 (satisfied) to 4 (dissatisfied). For all domains, a higher score indicates a more severe symptom burden or a greater negative impact on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Artur Biktimirov, MD, Study Chair — Federal Autonomous Educational Institution of Higher Education FEFU; Federal Center of Brain Research and Neurotechnologies; Mikhail Lebedev, PhD, Study Director — Faculty of Mechanics and Mathematics, Lomonosov Moscow State University; Daria Kleeva, Research Fellow, Principal Investigator — Vladimir Zelman Center for Neurobiology and Brain Rehabilitation, Skolkovo Institute of Science and Technology; Alexander Kaplan, D.Sci., Ph.D., Study Director — Faculty of Biology, Lomonosov Moscow State University
Locations (3):
- Russia (3):
  - Federal Autonomous Educational Institution of Higher Education FEFU, Vladivostok, Primorskiy (Maritime) Kray
  - Federal Center of Brain Research and Neurotechnologies, Moscow
  - Vladimir Zelman Center for Neurobiology and Brain Rehabilitation, Skolkovo Institute of Science and Technology, Moscow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith SE, Ma V, Gonzalez C, Chapman A, Printz D, Voytek B, Soltani M. Clinical EEG slowing induced by electroconvulsive therapy is better described by increased frontal aperiodic activity. Transl Psychiatry. 2023 Nov 16;13(1):348. doi: 10.1038/s41398-023-02634-9. PMID 37968263
- [Background] Simis M, Doruk Camsari D, Imamura M, Filippo TRM, Rubio De Souza D, Battistella LR, Fregni F. Electroencephalography as a Biomarker for Functional Recovery in Spinal Cord Injury Patients. Front Hum Neurosci. 2021 Apr 9;15:548558. doi: 10.3389/fnhum.2021.548558. eCollection 2021. PMID 33897390
- [Background] Jensen MP, Sherlin LH, Gertz KJ, Braden AL, Kupper AE, Gianas A, Howe JD, Hakimian S. Brain EEG activity correlates of chronic pain in persons with spinal cord injury: clinical implications. Spinal Cord. 2013 Jan;51(1):55-8. doi: 10.1038/sc.2012.84. Epub 2012 Jul 17. PMID 22801188
- [Background] Lopez-Larraz E, Montesano L, Gil-Agudo A, Minguez J, Oliviero A. Evolution of EEG Motor Rhythms after Spinal Cord Injury: A Longitudinal Study. PLoS One. 2015 Jul 15;10(7):e0131759. doi: 10.1371/journal.pone.0131759. eCollection 2015. PMID 26177457